CLINICAL TRIAL: NCT04570657
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of MEDI3506 in Adult Participants With Uncontrolled Moderate-to-severe Asthma
Brief Title: Study to Assess the Efficacy and Safety of MEDI3506 in Adults With Uncontrolled Moderate-to-severe Asthma
Acronym: FRONTIER-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9181C00001; 140910 (Other: FDA); 2020-000789-40 (EudraCT Number)
Record Dates: First submitted 2020-08-07; First posted 2020-09-30 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: MEDI3506; lung function; IL-33; inflammation
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI3506 Dose 1 (Experimental): Approximately 76 participants will be randomized to this arm to receive the higher dose of MEDI3506
  Interventions: Biological: MEDI3506
- MEDI3506 Dose 2 (Experimental): Approximately 76 participants will be randomized to this arm to receive the lower dose of MEDI3506
  Interventions: Biological: MEDI3506
- Placebo (Placebo Comparator): Approximately 76 participants will be randomized to this arm. Participants in this group will receive the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MEDI3506 — Participants will receive multiple doses of MEDI3506 at dose level 1 or dose level 2
  Arms: MEDI3506 Dose 1; MEDI3506 Dose 2
Drug: Placebo — Participants will receive multiple doses of placebo
  Arms: Placebo

SUMMARY:
Study D9181C00001 is a Phase II, randomised, double-blind, placebo-controlled, parallel group, proof of concept study to evaluate the efficacy, safety, pharmacokinetics (PK) and immunogenicity of MEDI3506 in adult participants with uncontrolled moderate to severe asthma on standard of care (SOC). Up to approximately 80 sites globally will participate in this study.

Approximately 228 participants will be randomized to 3 treatment groups in a 1:1:1 ratio to receive MEDI3506 dose 1, MEDI3506 dose 2, or placebo.

ELIGIBILITY:
INCLUSION CRITERIA

* Aged 18 to < 65 years of age
* Physician-diagnosed asthma of early onset, defined as development of asthma before the age of 25 years.
* History of ≥ 1 asthma exacerbation in previous 24 months
* Treated with medium to high dose ICS defined as total daily dose of > 250 g fluticasone dry powder or equivalent, for at least 12 months and on a stable dose for ≥ 3 months.
* Stable LABA therapy for ≥ 3 months.
* An ACQ-6 score ≥ 1.5.
* Morning pre-BD FEV1 ≥ 40% predicted normal and > 1 L.
* Morning pre-BD FEV1 < 85% predicted normal.
* Participants with documented evidence of asthma as demonstrated by either:
* BD reversibility, within 12 months, or at screening, or
* Positive methacholine challenge test within 12 months.
* Bodyweight ≥ 40 kg and BMI < 40 kg/m2.
* For female participants, a negative pregnancy test.
* Abide by contraception requirements for males and females
* Provide informed consent

EXCLUSION CRITERIA

* Participants with a positive diagnostic nucleic acid test for SARS-CoV-2.
* Participants with a significant COVID-19 illness within 6 months of enrolment:
* Participants with a recent history of, or who have a positive test for, infective hepatitis or unexplained jaundice, or participants who have been treated for hepatitis B, hepatitis C, or HIV.
* Evidence of active or latent TB:
* An LVEF < 45% measured by echocardiogram during screening.
* A family history of heart failure.
* Current smokers or recent ex-smokers i.e., have quit e cigarettes or other inhaled tobacco products ≤ 6 months prior to SV1.
* Ex-smokers with a total smoking history of > 10 pack years.
* As judged by the investigator, any evidence of any active medical or psychiatric condition or other reason (prior to randomisation) that in the investigator's opinion makes it undesirable for the participant to participate in the study.
* Any clinically important pulmonary disease other than asthma.
* Any other clinically relevant abnormal findings on physical examination or laboratory testing, that in the opinion of the investigator or medical monitor might compromise the safety of the participant in the study or interfere with evaluation of the study intervention.
* A known history of severe reaction to any medication including biologic agents or human gamma globulin therapy.
* History of, or a reason to believe, a participant has a history of, drug or alcohol abuse within the past 2 years.
* Current diagnosis of cancer.
* History of cancer, except if treated with apparent success with curative therapy (response duration of > 5 years).
* History of allogeneic bone marrow transplant.
* A helminth parasitic infection diagnosed within 6 months prior to SV4 (randomisation) that has not been treated, or has not responded to SOC therapy.
* An asthma exacerbation within 8 weeks.
* Receiving any prohibited concomitant medications or therapies as specified in the protocol:

Known history of allergy or reaction to any component of the study intervention formulation, including hereditary fructose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (9):
  - Research Site, Bakersfield, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Coral Gables, Florida
  - Research Site, Ames, Iowa
  - Research Site, Missoula, Montana
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Boerne, Texas
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Godoy Cruz
  - Research Site, Lanús Este
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Germany (12):
  - Research Site, Berlin
  - Research Site, Cottbus
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Koblenz
  - Research Site, Landsberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Peine
  - Research Site, Schwerin
- Hungary (5):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Gödöllő
  - Research Site, Százhalombatta
  - Research Site, Szeged
- Poland (10):
  - Research Site, Bialystok
  - Research Site, Bychawa
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Tarnów
  - Research Site, Wroclaw
- South Africa (8):
  - Research Site, Bellville
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pretoria
  - Research Site, Welkom
- United Kingdom (4):
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, High Wycombe
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: d9181c00001-study-synopsis_Redacted_pdfA.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9181C00001&attachmentIdentifier=ad9f60d8-283b-41ff-808d-263adeba65f9&fileName=d9181c00001-study-synopsis_Redacted_pdfA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and randomised in 52 study centres in 7 countries including Argentina, Germany, Hungary, Poland, South Africa, the United Kingdom, and the United States from 17 September 2020. The last participant completed their last study visit on 06 February 2023.
Pre-assignment Details: Adult participants with uncontrolled moderate to severe asthma were randomised in a 1:1:1 ratio to receive tozorakimab (MEDI3506) Dose A (lower dose), tozorakimab Dose B (higher dose), or placebo. Of the 478 participants screened, 250 were enrolled, and of these, 15 were excluded from analysis due to invalidity of data (see limitations and caveats for further details).
Groups:
- Tozorakimab Dose A: Participants were randomised to receive tozorakimab Dose A by subcutaneous (SC) injection.
- Tozorakimab Dose B: Participants were randomised to receive tozorakimab Dose B by SC injection.
- Placebo: Participants were randomised to receive placebo by SC injection.
Period: Overall Study
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Started | 77 | 77 | 81
Intent to Treat (ITT) Population | 77 | 77 | 81
As-treated Population | 77 | 77 | 81
Pharmacokinetic (PK) Population | 75 | 77 | 0
Completed | 76 | 74 | 77
Not Completed | 1 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo | Total
Number analyzed (Participants) | 77 | 77 | 81 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.97) | 43.1 (12.37) | 48.3 (10.41) | 44.5 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 43 | 150
  Male | 24 | 23 | 38 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 24 | 33 | 83
  Not Hispanic or Latino | 51 | 53 | 48 | 152
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 4 | 8 | 7 | 19
  White | 71 | 67 | 72 | 210
  Other | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Pre-bronchodilator (Pre-BD) Forced Expiratory Volume in the First Second (FEV1) as Measured in the Study Clinic
Description: In-clinic spirometry measurements were taken prior to the administration of bronchodilators. Baseline was the last measurement prior to first injection of investigational product (IP).
  The least squares (LS) means, LS mean differences and 80% confidence intervals (CIs), and one-sided p-value results were based on a mixed model repeated measures (MMRM). The model included fixed effects for baseline, background medication, geographic region, baseline inhaled corticosteroids (ICS) total daily dose, visit, treatment, and the baseline by visit and treatment by visit interactions. Visits within participant were considered as repeated measurements.
Time Frame: Baseline and week 16
Population: The ITT population included participants who were randomised and received any study intervention. Participants with data available are included.
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 76 | 77 | 81
litres | 0.148 (0.047) | 0.116 (0.048) | 0.112 (0.046)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.267, MMRM — One-sided p-value; LS mean difference = 0.036, 80% CI 2-sided [-0.038 to 0.111] — Tozorakimab Dose A - Placebo
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.473, MMRM — One-sided p-value; LS mean difference = 0.004, 80% CI 2-sided [-0.071 to 0.079] — Tozorakimab Dose B - Placebo

2. Secondary Outcome: Change From Baseline to Weeks 8 and 16 in Post-bronchodilator (Post-BD) FEV1 as Measured in the Study Clinic
Description: In-clinic spirometry measurements were taken following the use of bronchodilators. Bronchodilatation was induced using albuterol (90 µg metered dose), salbutamol (100 µg metered dose), or levalbuterol (45 µg metered dose), and measurements were taken after up to a maximum of 4 inhalations. Baseline was the last measurement prior to first injection of IP.
  The LS means, LS mean differences and 80% CIs, and one-sided p-value results were based on MMRM. The model included fixed effects for baseline, background medication, geographic region, baseline ICS total daily dose, visit, treatment, and the baseline by visit and treatment by visit interactions. Visits within participant were considered as repeated measurements.
Time Frame: Baseline and weeks 8 and 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 24 | 25 | 35
litres
  Week 8 | -0.062 (0.067) | 0.008 (0.068) | -0.050 (0.060)
  Week 16 | -0.064 (0.067) | -0.050 (0.068) | -0.026 (0.060)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.437, MMRM — One-sided p-value; LS mean difference = -0.012, 80% CI 2-sided [-0.110 to 0.086] — Week 8: Tozorakimab Dose A - Placebo
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.221, MMRM — One-sided p-value; LS mean difference = 0.059, 80% CI 2-sided [-0.039 to 0.157] — Week 8: Tozorakimab Dose B - Placebo
Statistical Analysis 3: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.308, MMRM — One-sided p-value; LS mean difference = -0.038, 80% CI 2-sided [-0.136 to 0.060] — Week 16: Tozorakimab Dose A - Placebo
Statistical Analysis 4: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.372, MMRM — One-sided p-value; LS mean difference = -0.025, 80% CI 2-sided [-0.122 to 0.072] — Week 16: Tozorakimab Dose B - Placebo

3. Secondary Outcome: Serum Concentrations of Tozorakimab
Description: Tozorakimab serum concentrations were measured using a validated assay method.
Time Frame: Pharmacokinetic (PK) samples were taken pre-dose (day 1) and at weeks 1, 4, 8, 12, 16, 20, and 24
Population: The PK population included participants who received at least one dose of tozorakimab and had at least one detectable serum concentration measurement post-first dose of study intervention. Participants with data available at each time point are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B
Number analyzed (Participants) | 75 | 77
µg/L
  Pre-dose: number analyzed (Participants) | 74 | 77
  Pre-dose | NA (NA) — Geometric mean (CV%) could not be calculated due to too many samples with tozorakimab concentrations below the limit of quantification. | NA (NA) — Geometric mean (CV%) could not be calculated due to too many samples with tozorakimab concentrations below the limit of quantification.
  Week 1: number analyzed (Participants) | 74 | 76
  Week 1 | 8939.24 (367.31) | 18374.15 (239.89)
  Week 4: number analyzed (Participants) | 72 | 72
  Week 4 | 2165.82 (180.17) | 4102.04 (168.60)
  Week 8: number analyzed (Participants) | 74 | 70
  Week 8 | 2680.07 (113.59) | 4476.11 (109.27)
  Week 12: number analyzed (Participants) | 74 | 75
  Week 12 | 2673.94 (121.08) | 4646.57 (153.62)
  Week 16: number analyzed (Participants) | 71 | 72
  Week 16 | 2742.93 (128.83) | 5007.93 (117.76)
  Week 20: number analyzed (Participants) | 75 | 72
  Week 20 | 356.56 (177.25) | 761.75 (152.78)
  Week 24: number analyzed (Participants) | 74 | 72
  Week 24 | 80.36 (170.34) | 146.67 (214.16)

4. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Description: ADA prevalence is the number of participants ADA positive (ADA+) at baseline and/or post-baseline. Treatment-emergent ADA+ (TE-ADA +) positive is defined as being either of treatment-induced ADA+ (ADA negative [ADA-] at baseline and at least one post-baseline ADA+) and treatment-boosted ADA+ (ADA+ at baseline and baseline titre is boosted by ≥ 4-fold increase at ≥ 1 post-baseline time point). Treatment-emergent ADA- (TE-ADA-) is defined as ADA+ but not fulfilling the definition of TE-ADA+. ADA persistently positive is defined as ADA- at baseline and ADA+ at ≥ 2 post-baseline assessment with ≥ 16 weeks between first and last positive assessments, or ADA+ at the last post-baseline assessment. ADA transiently positive is defined as ADA- at baseline, having at least one post-baseline ADA+ assessment and not fulfilling the conditions of ADA persistently positive. Baseline is defined as the last ADA assessment prior to first injection of IP.
Time Frame: Blood samples were taken pre-dose (day 1) and at weeks 1, 4, 8, 12, 16, and 24
Population: The as-treated population included participants who were randomised and received any study intervention. Participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 77 | 77 | 81
Participants
  ADA prevalence | 3 | 3 | 1
  TE-ADA+: number analyzed (Participants) | 75 | 77 | 81
  TE-ADA+ | 3 | 2 | 1
  Treatment-induced ADA+: number analyzed (Participants) | 75 | 77 | 81
  Treatment-induced ADA+ | 3 | 2 | 1
  TE-ADA-: number analyzed (Participants) | 75 | 77 | 81
  TE-ADA- | 0 | 1 | 0
  Both baseline and post-baseline positive: number analyzed (Participants) | 74 | 77 | 81
  Both baseline and post-baseline positive | 0 | 1 | 0
  ADA persistently positive: number analyzed (Participants) | 74 | 77 | 81
  ADA persistently positive | 3 | 1 | 0
  ADA transiently positive: number analyzed (Participants) | 74 | 77 | 81
  ADA transiently positive | 0 | 1 | 1

5. Secondary Outcome: Change From Baseline to Week 16 in the Asthma Control Questionnaire-6 (ACQ-6) Score
Description: In the ACQ-6, participants were asked to recall how their asthma has been during the previous week by responding to one BD-use question and 5 symptom questions. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between >0.75 and <1.5 indicate partly controlled asthma, and scores ≥1.5 indicate not well-controlled asthma. Results were based on an MMRM which included fixed effects for baseline, background medication, geographic region, baseline ICS total daily dose, visit, treatment and the baseline by visit and treatment by visit interactions. Visits within participant were considered as repeated measurements. A negative change from baseline indicates an improvement in asthma control.
Time Frame: Baseline and week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 76 | 77 | 81
score on a scale | -0.925 (0.117) | -0.942 (0.117) | -0.895 (0.112)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.416, MMRM — One-sided p-value; LS mean difference = -0.030, 80% CI 2-sided [-0.215 to 0.154] — Tozorakimab Dose A - Placebo
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.371, MMRM — One-sided p-value; LS mean difference = -0.047, 80% CI 2-sided [-0.231 to 0.137] — Tozorakimab Dose B - Placebo

6. Secondary Outcome: Number of Participants With a Decrease in ACQ-6 Score ≥ 0.5 From Baseline to Week 16
Description: In the ACQ-6, participants were asked to recall how their asthma has been during the previous week by responding to one BD-use question and 5 symptom questions. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between >0.75 and <1.5 indicate partly controlled asthma, and scores ≥1.5 indicate not well-controlled asthma. A decrease in ACQ-6 score baseline indicates an improvement in asthma control, and individual changes of at least 0.5 are considered clinically meaningful.
Time Frame: Baseline and week 16
Population: The ITT population included participants who were randomised and received any study intervention. Participants with evaluable ACQ-6 scores were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 73 | 74 | 77
Participants | 53 | 56 | 53
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.612, Chi-squared; Odds Ratio (OR) = 1.20, 80% CI 2-sided [0.76 to 1.90]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.348, Chi-squared; Odds Ratio (OR) = 1.41, 80% CI 2-sided [0.88 to 2.25]

7. Secondary Outcome: Number of Participants Achieving ACQ-6 Well Controlled Status at Week 16
Description: In the ACQ-6, participants were asked to recall how their asthma has been during the previous week by responding to one BD-use question and 5 symptom questions. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between >0.75 and <1.5 indicate partly controlled asthma, and scores ≥1.5 indicate not well-controlled asthma.
Time Frame: Baseline and week 16
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 73 | 74 | 77
Participants | 17 | 18 | 21
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.575, Chi-squared; Odds Ratio (OR) = 0.81, 80% CI 2-sided [0.50 to 1.31]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.679, Chi-squared; Odds Ratio (OR) = 0.86, 80% CI 2-sided [0.53 to 1.38]

8. Secondary Outcome: Change From Baseline to Week 16 in St George's Respiratory Questionnaire (SGRQ) Domain and Total Scores
Description: The SGRQ is a 50-item patient-reported outcome instrument to measure the health status of participants with airway obstruction diseases, giving a total score and 3 domain scores (symptoms, activity, and impacts). The total score is expressed as a percentage of overall impairment, with 100 representing the worst possible health status and 0 the best possible health status. Each domain score ranges from 0 to 100, with higher scores indicating greater impairment. A negative change from baseline indicates an improvement in impairments. Results were based on an MMRM which included fixed effects for baseline, background medication, geographic region, baseline ICS total daily dose, visit, treatment and the baseline by visit and treatment by visit interactions. Visits within participant were considered as repeated measurements.
Time Frame: Baseline and week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 76 | 77 | 80
score on a scale
  SGRQ Activity Total Score | -10.340 (2.477) | -11.706 (2.507) | -10.342 (2.390)
  SGRQ Impacts Total Score | -8.237 (1.750) | -8.509 (1.774) | -6.816 (1.689)
  SGRQ Symptoms Total Score | -15.290 (2.828) | -19.130 (2.873) | -15.981 (2.726)
  SGRQ Total Score | -10.133 (1.815) | -11.366 (1.838) | -9.470 (1.750)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.500, MMRM — One-sided p-value; LS mean difference = 0.002, 80% CI 2-sided [-3.825 to 3.828] — SGRQ Activity Total Score: Tozorakimab Dose A - Placebo
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.324, MMRM — One-sided p-value; LS mean difference = -1.364, 80% CI 2-sided [-5.198 to 2.470] — SGRQ Activity Total Score: Tozorakimab Dose B - Placebo
Statistical Analysis 3: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.248, MMRM — One-sided p-value; LS mean difference = -1.421, 80% CI 2-sided [-4.103 to 1.260] — SGRQ Impacts Total Score: Tozorakimab Dose A - Placebo
Statistical Analysis 4: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.210, MMRM — One-sided p-value; LS mean difference = -1.694, 80% CI 2-sided [-4.383 to 0.996] — SGRQ Impacts Total Score: Tozorakimab Dose B - Placebo
Statistical Analysis 5: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.420, MMRM — One-sided p-value; LS mean difference = 0.691, 80% CI 2-sided [-3.715 to 5.096] — SGRQ Symptoms Total Score: Tozorakimab Dose A - Placebo
Statistical Analysis 6: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.181, MMRM — One-sided p-value; LS mean difference = -3.150, 80% CI 2-sided [-7.579 to 1.280] — SGRQ Symptoms Total Score: Tozorakimab Dose B - Placebo
Statistical Analysis 7: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.380, MMRM — One-sided p-value; LS mean difference = -0.663, 80% CI 2-sided [-3.454 to 2.129] — SGRQ Total Score: Tozorakimab Dose A - Placebo
Statistical Analysis 8: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.192, MMRM — One-sided p-value; LS mean difference = -1.896, 80% CI 2-sided [-4.694 to 0.903] — SGRQ Total Score: Tozorakimab Dose B - Placebo

9. Secondary Outcome: Number of Participants With a Decrease in SGRQ Total Score of ≥ 4 Points From Baseline to Week 16
Description: The SGRQ is a 50-item patient-reported outcome instrument to measure the health status of participants with airway obstruction diseases, giving a total score and 3 domain scores (symptoms, activity, and impacts). The total score is expressed as a percentage of overall impairment, with 100 representing the worst possible health status and 0 the best possible health status. A decrease in the SGRQ total score indicates an improvement in overall impairment.
Time Frame: Baseline and week 16
Population: The ITT population included participants who were randomised and received any study intervention. Participants with evaluable SGRQ scores were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 73 | 74 | 77
Participants | 50 | 53 | 54
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.828, Chi-squared; Odds Ratio (OR) = 0.93, 80% CI 2-sided [0.59 to 1.46]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.840, Chi-squared; Odds Ratio (OR) = 1.07, 80% CI 2-sided [0.68 to 1.70]

10. Secondary Outcome: Number of Participants With at Least One Asthma CompEx Event From Baseline to Week 16
Description: Asthma CompEx is a combination of exacerbations of asthma and diary events (i.e., a combination of electronic diary [eDiary] variables). eDiary events are defined by criteria using morning/evening diary variables of PEF, symptoms, and use of rescue medication. A participant was considered to have a CompEx event if they had one or both of an asthma exacerbation or diary event. For participants who did not experience an on-treatment CompEx event, date of censoring was the minimum between the date of last dose + 28 days, and the last day of eDiary recording during the on-treatment period.
Time Frame: Baseline to week 16
Population: The ITT population included participant who were randomised and received any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 77 | 77 | 81
Participants | 19 | 15 | 15
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.239, Regression, Cox — One-sided p-value; Cox regression model with treatment group, background medication, geographic region, and ICS total daily dose as covariates; Hazard Ratio (HR) = 1.3, 80% CI 2-sided [0.8 to 2.0]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.461, Regression, Cox — One-sided p-value; [statistical method as in outcome 10, analysis 1]; Hazard Ratio (HR) = 1.0, 80% CI 2-sided [0.6 to 1.7]

11. Secondary Outcome: Asthma CompEx Annualised Event Rate
Description: The annualised rate of asthma CompEx events was calculated as the total number of asthma CompEx events / (date of last dose of IP + 28 - date of first dose of IP - recovery time + 1) / 365.25.
  The rates, rate ratios, and one-sided p-values were estimated from a negative binomial regression, with the log(follow up time) included as an offset term. The dependent variable will be the number of CompEx events during the on-treatment period (i.e., from baseline to last dose date +28 days), and the model will include treatment group, background medication, geographic region and baseline ICS total daily dose as covariates.
Time Frame: Baseline to week 16
Population: The ITT population included participants who were randomised and received any study intervention.
Measure: Number (80% Confidence Interval); unit: events per participant-treatment year
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 77 | 77 | 81
events per participant-treatment year | 0.86 [0.58 to 1.28] | 0.69 [0.44 to 1.07] | 0.99 [0.68 to 1.44]
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.346, Negative binomial regression — One-sided p-value; Rate ratio = 0.87, 80% CI 2-sided [0.56 to 1.36]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.166, Negative binomial regression — One-sided p-value; Rate ratio = 0.70, 80% CI 2-sided [0.43 to 1.12]

12. Secondary Outcome: Percent Change From Baseline to Week 16 in Concentration of Fractional Exhaled Nitric Oxide (FeNO) in Exhaled Breath
Description: A standardised single-breath FeNO test was performed to evaluate airway inflammation. Results were based on MMRM on log-transformed change from baseline. Log-transformed change from baseline is calculated as the visit value in log minus the baseline value in log. The results from the model were then back transformed. The model included fixed effects for baseline (in log), background medication, geographic region, baseline ICS total daily dose, visit, treatment and the baseline by visit and treatment by visit interactions. Visits within subject were considered as repeated measurements.
Time Frame: Baseline and week 16
Population: as for outcome 1
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: percent change
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 74 | 77 | 81
percent change | -17.429 [-23.423 to -10.965] | -16.500 [-22.548 to -9.981] | -5.007 [-11.612 to 2.091]
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Test type: Superiority; p = 0.029, MMRM — One-sided p-value; Geometric LS mean ratio = 0.869, 80% CI 2-sided [0.791 to 0.956]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; Test type: Superiority; p = 0.040, MMRM — One-sided p-value; Geometric LS mean ratio = 0.879, 80% CI 2-sided [0.800 to 0.966]

13. Other Pre Specified Outcome: Change From Baseline to Week 16 in Pre-BD FEV1 as Measured in the Study Clinic: Analysis Per Number of Exacerbations in Last 12 Months
Description: In-clinic spirometry measurements were taken prior to the administration of bronchodilators. Baseline was the last measurement prior to first injection of IP.
  The LS means, LS mean differences and 80% CIs, and one-sided p-value results were based on MMRM. The model included fixed effects for baseline, visit, treatment, and the baseline by visit and treatment by visit interactions. Visits within participant were considered as repeated measurements. Analysis is presented by the number of asthma exacerbations experienced within the 12 months prior to baseline (1 or ≥ 2 exacerbations in the previous 12 months).
Time Frame: Baseline and week 16
Population: Participants in the ITT population with 1 or ≥ 2 exacerbations in the previous 12 months are included in the analysis. The ITT population included participants who were randomised and received any study intervention. Participants with data available are included.
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 45 | 47 | 52
litres
  1 Exacerbation in Last 12 Months | 0.188 (0.065) | 0.042 (0.070) | 0.165 (0.062)
  ≥ 2 Exacerbations in Last 12 Months: number analyzed (Participants) | 31 | 30 | 29
  ≥ 2 Exacerbations in Last 12 Months | 0.059 (0.067) | 0.194 (0.065) | -0.018 (0.069)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; 1 Exacerbation in Last 12 Months; Test type: Superiority; p = 0.385, MMRM — One-sided p-value; alpha = 0.1; LS mean difference = 0.023, 80% CI 2-sided [-0.078 to 0.124] — Tozorakimab Dose A - Placebo
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; 1 Exacerbation in Last 12 Months; Test type: Superiority; p = 0.060, MMRM — One-sided p-value; alpha = 0.1; LS mean difference = -0.123, 80% CI 2-sided [-0.224 to -0.022] — Tozorakimab Dose B - Placebo
Statistical Analysis 3: Comparison: Tozorakimab Dose A vs Placebo; ≥ 2 Exacerbation in Last 12 Months; Test type: Superiority; p = 0.186, MMRM — One-sided p-value; alpha = 0.1; LS mean Difference = 0.077, 80% CI 2-sided [-0.034 to 0.187] — Tozorakimab Dose A - Placebo
Statistical Analysis 4: Comparison: Tozorakimab Dose B vs Placebo; ≥ 2 Exacerbation in Last 12 Months; Test type: Superiority; p = 0.007, MMRM — One-sided p-value; alpha = 0.1; LS mean difference = 0.212, 80% CI 2-sided [0.102 to 0.322] — Tozorakimab Dose B - Placebo

14. Other Pre Specified Outcome: Eosinophil Count
Description: The eosinophil count at baseline and week 16 are presented. Baseline was defined as the last measurement prior to first injection of IP.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^9 cells/L
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
Number analyzed (Participants) | 77 | 77 | 81
10^9 cells/L
  Baseline | 0.187 (80.4) | 0.200 (88.4) | 0.178 (83.3)
  Week 16: number analyzed (Participants) | 65 | 70 | 73
  Week 16 | 0.122 (82.9) | 0.136 (77.6) | 0.185 (93.2)
Statistical Analysis 1: Comparison: Tozorakimab Dose A vs Placebo; Analysis at Week 16 based on MMRM which included fixed effects for baseline, background medication, geographic region, baseline ICS total daily dose, visit, treatment and the baseline by visit and treatment by visit interactions; Test type: Superiority; p < 0.001, MMRM — One-sided p-value; Geometric LS Mean Ratio = 0.630, 80% CI 2-sided [0.559 to 0.710]
Statistical Analysis 2: Comparison: Tozorakimab Dose B vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, MMRM — One-sided p-value; Geometric LS Mean Ratio = 0.675, 80% CI 2-sided [0.599 to 0.760]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24 (up to 24 weeks)
Arm/Group | Tozorakimab Dose A | Tozorakimab Dose B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/77 | 4/77 | 2/81
Other Adverse Events (participants affected / at risk) | 25/77 | 20/77 | 20/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tozorakimab Dose A (N=77) | Tozorakimab Dose B (N=77) | Placebo (N=81)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tozorakimab Dose A (N=77) | Tozorakimab Dose B (N=77) | Placebo (N=81)
COVID-19 (Infections and infestations) | 15 (17) | 10 (12) | 11 (12)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (6) | 4 (5)
Injection site erythema (General disorders) | 4 (5) | 7 (15) | 2 (5)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Injection site swelling (General disorders) | 0 (0) | 4 (5) | 1 (4)
Injection site urticaria (General disorders) | 1 (1) | 4 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
15 participants enrolled at 1 study centre were excluded from the final analysis due to inability to confirm the validity of the data reported by the site. The exclusion of data from this site did not change the interpretation of the primary endpoint, or results in a significant change to the interpretation of any other endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT04570657/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04570657/SAP_001.pdf